CLINICAL TRIAL: NCT06602856
Title: The Benefits of Pre-hospital POCUS Examinations in Air Rescue
Brief Title: Point-of-care-ultrasound in Swiss Air Rescue Rega
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-01154
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Point-of-care-ultrasound; Emergency Treatment
Keywords: POCUS; Helicopter emergency medical service; Diagnostic quality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Point-of-care ultrasound examination — We are investigating the extent to which pre-hospital point-of-care ultrasound examination influences the further deployment tactics, medical treatment and choice of destination hospital for patients.

SUMMARY:
The aim of the study is, on the one hand, to objectively investigate the patient-oriented benefits of prehospital point-of-care ultrasound (POCUS) examinations under the conditions of the helicopter emergency medical services (HEMS) in Switzerland. On the other hand, the study will show what the diagnostic quality of prehospital POCUS examinations is and how emergency medical teams can be trained to use POCUS in the future.

HEMS crew members will answer a short online questionaire about how findings of their POCUS examination has influenced their medical treatment, diagnosis and selection of target hospital for the patient (primary outcome parameters).

In addition, a study nurse will query the findings of the in-hospital diagnostic tests and compare them with the findings of the pre-hospital POCUS examination. This will enable the investigators to evaluate the diagnostic quality of the prehospital POCUS examination and to identify which findings are often not recognised in the POCUS. The subjective satisfaction and assessment of the benefit of the POCUS examination by the respective users will also be recorded (secondary outcome parameters).

ELIGIBILITY:
Inclusion Criteria:

* All patients in whom the treating Rega team uses POCUS pre-hospital
* existing written General Consent (with permission to use patient data for research)

Exclusion Criteria:

* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Swiss Air Rescue Rega treats more than 12,000 patients annually. It is estimated that 1,000 of these will undergo a prehospital POCUS examination. These include both trauma patients and patients with medical diseases such as pulmonary oedema, COPD, myocardial infarction, etc.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis | During HEMS mission, estimated to be on average of 30-60 minutes
  Number of patients and clinical pictures/injuries of patients in whom the findings of prehospital POCUS influenced the further course of action with regard to diagnosis?
Therapeutic interventions | During HEMS mission, estimated to be on average 30-60 minutes
  Number of patients and clinical pictures/injuries of patients in whom the findings of prehospital POCUS influenced the further course of action with regard to therapeutic interventions (e.g. pleural decompression, fluid therapy, medication)?
Transportation target | During HEMS mission, estimated to be on average 30-60 minutes
  Number of patients and clinical pictures/injuries of patients in whom the findings of prehospital POCUS influenced the further course of action with regard to selection of the target hospital

SECONDARY OUTCOMES:
Missed findings | 1 day
  Number of findings and which findings are missed during prehospital POCUS?
Users' subjective assessment | 1 day
  Personal assessment of the users with regard to the benefit for the patient and the applicability of prehospital POCUS on a numeric rating scale from 1 to 10 (1=no benefit, 10=maximum benefit)
Diagnostic quality | 1 day
  Interrater reliability analysis with the target size Cohen's kappa between POCUS findings and findings of in-hospital imaging (ultrasound, conventional X-ray, computed tomography)?

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Knapp, Dr., Principal Investigator — Bern University Hospital
Locations (1):
- Swiss Air Rescue Rega, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided